CLINICAL TRIAL: NCT03558035
Title: New Strategy of Improving Treatment Outcome and Larynx-preservation Rate in Locally Advanced Hypopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun-Lin Yi, MD, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC2014L12
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Hypopharyngeal Cancer
Keywords: Hypopharyngeal carcinoma; Locally advanced; Multi-disciplinary treatment; Functional Magnetic Resonance Imaging; Prognosis
MeSH Terms: conditions — Hypopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction chemotherapy and concurret chemoradiotherapy group (Experimental): Patients receive 2 cycles of paclitaxel, cisplatin and 5-Fluorouracil chemotherapy followed by Surgery or Chemo-radiotherapy according to the response status after induction chemo.
  Interventions: Drug: Induction CT+ CRT group
- Concurrent chemoradiotherapy group (Active Comparator): Patients receive single-agent cisplatin chemotherapy concurrent with Radiotherapy
  Interventions: Radiation: Concurrent CRT group

INTERVENTIONS:
Drug: Induction CT+ CRT group — Induction CT: Paclitaxel 175mg/m2 IV on d1 and d22, cisplatin 75mg/m2 IV on d1 and d22, 5-Fluorouracil 750mg/m2 IV continuously on d1-4 and d22-25, CRT: cisplatin 80mg/m2 IV on d1 of each 21 days cycle and 70 Gy radiotherapy
  Arms: Induction chemotherapy and concurret chemoradiotherapy group
Radiation: Concurrent CRT group — cisplatin 100mg/m2 IV on d1 of each 21 days cycle and 70 Gy radiotherapy
  Arms: Concurrent chemoradiotherapy group

SUMMARY:
To develope stratification treatment for the patients who have locally advanced hypopharyngeal carcinoma. Experimental group patients were treated individually according to the response status after induction chemotherapy, receiving chemoradiotherapy or surgery. Thus to achieve a better survival rate and a higher larynx-preservation rate as well as a lower treatment related toxicity rate compared with standard treatment.

DETAILED DESCRIPTION:
Eligiblity patient were assign to induction chemotherapy plus concurrent chemotherapy group (IC +CCRT group, Arm A)and concurrent chemoradiotherapy group(CCRT group, Arm B). For patients in Arm A, treatment response were evaluated after 2cycles, if the response reached partial response/complete response, patients received concurrent chemoradiotherapy, otherwise, patients will received surgery and radiotherpay/concurrent chemoradiotherapy after surgery. For patients received concurrent chemoradiotherapy (both in Arm A and Arm B) , treatment response were evaluated at 50 Gy. if response reached complete response or major partial response(>80% tumor regression), patients will received radical chemoradiotherapy, otherwise, patients will received surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of hypopharynx
* Stage III/IV M0, with T3/4 N0-3 or T1-4 N2-3
* Karnofsky Performance Status>=70
* Have measurable lesions on CT/MRI
* Treatment for the first time
* Expected lifetime > 6 months
* Normal blood test, hepatic and renal functions
* Normal hearing
* Can understand and sign the consent
* Have follow up condition

Exclusion Criteria:

* Past malignancies history (except for stage I non-melanoma skin cancer or cervical carcinoma in situ)
* Previously treatment for cancer
* Pregnant or breeding woman, female without contraception
* Enrolling in other drug trials
* Severe comorbidities including myocardial infarction, arrhythmia, cerebral vascular disease, ulceration disease, mental disease and uncontrolled diabetes
* Without follow up
* Receive target therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2014-09; Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
disease free survival | 5 year
distant-metastasis free survival | 5 year
larynx-preservation rate | 5 year
treatment related toxicities | 2 year
  hematology and surgery related complications

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, Professor, Principal Investigator — CAMS
Locations (1):
- Cancer hospital, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Blanchard P, Baujat B, Holostenco V, Bourredjem A, Baey C, Bourhis J, Pignon JP; MACH-CH Collaborative group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): a comprehensive analysis by tumour site. Radiother Oncol. 2011 Jul;100(1):33-40. doi: 10.1016/j.radonc.2011.05.036. Epub 2011 Jun 16. PMID 21684027
- [Background] Blanchard P, Bourhis J, Lacas B, Posner MR, Vermorken JB, Cruz Hernandez JJ, Bourredjem A, Calais G, Paccagnella A, Hitt R, Pignon JP; Meta-Analysis of Chemotherapy in Head and Neck Cancer, Induction Project, Collaborative Group. Taxane-cisplatin-fluorouracil as induction chemotherapy in locally advanced head and neck cancers: an individual patient data meta-analysis of the meta-analysis of chemotherapy in head and neck cancer group. J Clin Oncol. 2013 Aug 10;31(23):2854-60. doi: 10.1200/JCO.2012.47.7802. Epub 2013 Jul 8. PMID 23835714
- [Background] Pointreau Y, Garaud P, Chapet S, Sire C, Tuchais C, Tortochaux J, Faivre S, Guerrif S, Alfonsi M, Calais G. Randomized trial of induction chemotherapy with cisplatin and 5-fluorouracil with or without docetaxel for larynx preservation. J Natl Cancer Inst. 2009 Apr 1;101(7):498-506. doi: 10.1093/jnci/djp007. Epub 2009 Mar 24. PMID 19318632
- [Derived] Luo X, Huang X, Luo J, Xiao J, Wang K, Qu Y, Chen X, Zhang Y, Wu R, Wang J, Zhang J, Xu G, Gao L, Liu S, Wang X, He X, Luo D, Yi J. Induction TPF followed by concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locally advanced hypopharyngeal cancer: a preliminary analysis of a randomized phase 2 trial. BMC Cancer. 2022 Nov 29;22(1):1235. doi: 10.1186/s12885-022-10306-y. PMID 36447152